CLINICAL TRIAL: NCT00065767
Title: Cognitive and Neurophysiological Effects of Raloxifene in Alzheimer's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0049; 1R01AG029624-01 (NIH); IRB M1285
Record Dates: First submitted 2003-07-31; First posted 2003-08-04 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Postmenopausal women; Hormone therapy
MeSH Terms: conditions — Alzheimer Disease | interventions — Raloxifene Hydrochloride

INTERVENTIONS:
Drug: Raloxifene

SUMMARY:
The aim of this study is to determine the effectiveness of treatment with raloxifene, an estrogen-like medication approved by the Food and Drug Administration for the treatment of osteoporosis, in improving memory and the ability to live independently in postmenopausal women with Alzheimer's disease.

DETAILED DESCRIPTION:
The aim of this study is to determine the effectiveness of treatment with raloxifene, an estrogen-like medication (classified as Selective Estrogen Receptor Modulators (SER's)) approved by the Food and Drug Administration for the treatment of osteoporosis, in improving memory and the ability to live independently in postmenopausal women with Alzheimer's disease. Patients who volunteer for this study will need to visit the clinic 7 times (participate) over a period of five months and will receive either raloxifene or a harmless, inactive pill called a placebo. Neither the volunteers nor the study staff will know which type of pill a patient receives. Patients must be generally healthy and have mild-to-moderate dementia. There must be a patient caregiver who can watch for side effects and ensure that the patient takes the study pills on schedule over a period of three months.

Patients will undergo neuropsychological tests and an evaluation of the ability to live independently at each visit as well as laboratory evaluations, such as the taking of blood. Each visit will last approximately 3 hours. A total of 20 patients is being recruited to participate in this study at the University of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with Alzheimer's disease and without other dementias (diagnosed by study staff or from an outside clinic)
* Mini Mental Status Exam score greater than 15/30

Exclusion Criteria:

* History of deep vein thrombosis or blot clots
* Diabetes
* Active heart disease or stroke
* Liver problems including hepatitis
* Severe vision or hearing problems
* Tobacco use

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-09; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Asthana, MD, Principal Investigator — William S. Middleton VA Hospital, University of Wisconsin Memory Research Program
Locations (1):
- University of Wisconsin Memory Research Program, Madison, Wisconsin, United States

REFERENCES:
- [Background] Birge SJ, McEwen BS, Wise PM. Effects of estrogen deficiency on brain function. Implications for the treatment of postmenopausal women. Postgrad Med. 2001 Mar;Spec No:11-6. PMID 11296734
- [Background] Zec RF, Trivedi MA. The effects of estrogen replacement therapy on neuropsychological functioning in postmenopausal women with and without dementia: a critical and theoretical review. Neuropsychol Rev. 2002 Jun;12(2):65-109. doi: 10.1023/a:1016880127635. PMID 12371603
- [Background] Yaffe K. Estrogens, selective estrogen receptor modulators, and dementia: what is the evidence? Ann N Y Acad Sci. 2001 Dec;949:215-22. doi: 10.1111/j.1749-6632.2001.tb04024.x. PMID 11795356